CLINICAL TRIAL: NCT04187989
Title: Social Media Intervention for Cannabis Use in Emerging Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Erin Bonar, University of Michigan, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00152202; R34DA045712 (NIH)
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Results first posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Cannabis Use
Keywords: Social Media

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Media Intervention (Experimental): Facebook page that will deliver health information focused on increasing well-being and reducing risky behaviors.
  Interventions: Behavioral: Social Media Intervention
- Control (No Intervention): An Attention-Control E-News (control) condition

INTERVENTIONS:
Behavioral: Social Media Intervention — Information will be posted by e-coaches. You can interact with the e-coaches as well as other study members in your group.
  Arms: Social Media Intervention

SUMMARY:
The purpose of the study is to develop and test social media interventions to help young people increase well-being and reduce risky behaviors. The study will help researchers learn about ways to deliver wellness information in a way that is appealing and helpful to young people who use Facebook.

ELIGIBILITY:
Inclusion Criteria:

* self-report using cannabis at least 3 time per week or more often in the past month
* active Facebook profile
* view and click on a social media ad

Exclusion Criteria:

* fail identity verification based on 1) Internet Protocol (IP) addresses, 2) survey time completion, 3) repeat attempts, 4) survey responses, and 5) photo identification via a timestamped selfie sent to the research staff.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 149 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Bonar, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bonar EE, Goldstick JE, Chapman L, Bauermeister JA, Young SD, McAfee J, Walton MA. A social media intervention for cannabis use among emerging adults: Randomized controlled trial. Drug Alcohol Depend. 2022 Mar 1;232:109345. doi: 10.1016/j.drugalcdep.2022.109345. Epub 2022 Feb 3. PMID 35144238

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 2 waves of recruitment: Wave 1 (February 2020) occurred for participants residing in states without legal recreational cannabis; Wave 2 (May 2020) occurred for those living in states with legal recreational cannabis.
Period: Overall Study - 3-Month Follow-Up
Arm/Group | Social Media Intervention | Control
Started | 76 | 73
Completed (Completed 3-Month Follow-Up) | 70 | 65
Not Completed | 6 | 8
Not completed — Lost to Follow-up | 6 | 8
Period: Overall Study - 6-Month Follow-Up
Arm/Group | Social Media Intervention | Control
Started | 76 | 73
Completed (Completed 6-Month Follow-Up) | 68 | 65
Not Completed | 8 | 8
Not completed — Lost to Follow-up | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Social Media Intervention | Control | Total
Number analyzed (Participants) | 76 | 73 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.2 (2.3) | 20.9 (2.0) | 21.0 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 40 | 83
  Male | 33 | 33 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 56 | 69
  Not Hispanic or Latino | 63 | 17 | 80
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaska Native | 3 | 1 | 4
  Asian American | 3 | 4 | 7
  Black/African American | 8 | 7 | 15
  White | 42 | 43 | 85
  Multi-racial | 15 | 14 | 29
  Other race | 5 | 4 | 9
Total days of cannabis use in past 30 (from Timeline Follow Back: TLFB) [Mean (Standard Deviation); unit: days] | 20.8 (9.3) | 16.7 (11.1) | 18.8 (10.4)
Total estimated grams cannabis use from Timeline Follow Back (past 30 days) [Mean (Standard Deviation); unit: grams] — Population: 2 participants in the control group had missing baseline data on quantity
  grams
    number analyzed (Participants) | 76 | 71 | 147
    (all) | 21.5 (22.3) | 13.1 (17.6) | 17.5 (20.6)
Total consequences from Marijuana Adolescent Consequences Questionnaire [Mean (Standard Deviation); unit: count of consequences] — Population: 2 participants in the control group are missing data on the consequences measure
  count of consequences
    number analyzed (Participants) | 76 | 71 | 147
    (all) | 9.4 (4.8) | 10.1 (5.8) | 9.8 (5.3)
Perceived risk [Mean (Standard Deviation); unit: units on a scale] — Population: Two control participants were missing baseline data on this measure
  units on a scale
    number analyzed (Participants) | 76 | 71 | 147
    (all) | 3.1 (1.1) | 3.4 (1.1) | 3.2 (1.1)
Peer approval [Mean (Standard Deviation); unit: units on a scale] — Population: 3 control participants are missing data on this measure at baseline
  units on a scale
    number analyzed (Participants) | 76 | 70 | 146
    (all) | 1.0 (0.2) | 1.1 (0.3) | 1.05 (0.3)
Cannabis-impaired driving [Mean (Standard Deviation); unit: units on a scale] — Population: 2 control participants had missing data on this scale
  units on a scale
    number analyzed (Participants) | 76 | 71 | 147
    (all) | 11.1 (10.5) | 9.7 (8.8) | 10.4 (10.2)
Past 30-day other substance use index [Mean (Standard Deviation); unit: mid-point of range total score across 6] — Items from the Monitoring the Future Survey will be used to assess past 30 day use of 6 other substances - substances used and number of times of use. Response values will be summed for a total score using mid-point of the range scoring.
  Substances assessed include: hallucinogens, opioids, stimulants, sedatives, lsd, ecstasy
  Response scale:
  0 0 Occasions 1-2 Occasions 3-5 Occasions 6-9 Occasions 10-19 Occasions 20-39 Occasions 40 or More Occasions
  Higher scores = greater substance use
  mid-point of range total score across 6 | 2.0 (4.9) | 1.4 (3.6) | 1.70 (4.3)
Alcohol use days in past 30 (from Timeline Follow Back: TLFB) [Mean (Standard Deviation); unit: days] — Population: This measure restricted to only those participants who drank alcohol at baseline
  days
    number analyzed (Participants) | 59 | 43 | 102
    (all) | 6.2 (6.7) | 7.2 (7.2) | 6.6 (6.9)
Alcohol quantity (total drinks) in past 30 days [Mean (Standard Deviation); unit: estimated standard drinks] — Population: This measure restricted to those who drank alcohol at baseline.
  estimated standard drinks
    number analyzed (Participants) | 59 | 43 | 102
    (all) | 15.9 (15.6) | 17.4 (18.3) | 16.6 (16.7)

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Cannabis Use as Reported on the Timeline Follow-Back (TLFB)
Description: 30-day TLFB self-report will be used to assess total number of days of cannabis use.
Time Frame: 3-months post baseline
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Social Media Intervention | Control
Number analyzed (Participants) | 70 | 65
days | 18.0 (11.5) | 14.9 (11.7)
Statistical Analysis 1: Comparison: Social Media Intervention vs Control; We fixed linear mixed effects models adjusted for baseline values, balancing factors (age, sex, recreational cannabis), and included a random intercept for group because this is an individually randomized group treatment trial. We tested for treatment effects with a two-sided test of the coefficient for the treatment/control indicator, and estimated Cohen's D (mean difference between the 2 groups at follow-up divided by the total variation not captured by the fixed effects) along with 95% CIs; Test type: Other — Two-sided test of the null hypothesis of no difference between groups; p = .980, t-test, 2 sided; The p-value is for the coefficient of the treatment/control indicator in the above mixed model; Cohen's D = -.006, 95% CI 2-sided [-.478 to .466], Standard Error of Mean .239 — The effect size used is the adjusted Cohen's D, calculated from the coefficient for treatment group in the mixed model, divided by total pooled SD (the square root of the sum of the residual variance+the variance of the group-level random effects)

2. Primary Outcome: Frequency of Cannabis Use as Reported on the Timeline Follow-Back (TLFB)
Description: 30-day TLFB self-report will be used to assess total number of days of cannabis use.
Time Frame: 6-months post baseline
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Social Media Intervention | Control
Number analyzed (Participants) | 68 | 65
days | 16.8 (12.2) | 15.8 (11.8)
Statistical Analysis 1: Comparison: Social Media Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Other — Two-sided test of the null hypothesis of no difference between groups; p = .140, t-test, 2 sided — The p-value is for the coefficient of the treatment/control indicator in the above mixed model; Cohen's D = .265, 95% CI 2-sided [-.092 to .621], Standard Error of Mean .180 — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Quantity of Cannabis Used as Reported on the Timeline Follow-Back (TLFB)
Description: 30-day Timeline Follow-Back (TLFB) self-report will be used to assess quantity (grams) of cannabis consumed.
Time Frame: 3-months post baseline
Measure: Mean (Standard Deviation); unit: quantity (grams)
Arm/Group | Social Media Intervention | Control
Number analyzed (Participants) | 70 | 65
quantity (grams) | 19.8 (26.7) | 11.6 (15.6)

4. Primary Outcome: Quantity of Cannabis Used as Reported on the Timeline Follow-Back (TLFB)
Description: 30-day Timeline Follow-Back (TLFB) self-report will be used to assess quantity (grams) of cannabis consumed.
Time Frame: 6-months post baseline
Measure: Mean (Standard Deviation); unit: quantity (grams)
Arm/Group | Social Media Intervention | Control
Number analyzed (Participants) | 68 | 65
quantity (grams) | 15.5 (21.7) | 11.5 (15.0)
Statistical Analysis 1: Comparison: Social Media Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Other — Two-sided test of the null hypothesis of no difference between groups; p = .724, t-test, 2 sided — Two-sided test of the null hypothesis of no difference between groups; The p-value is for the coefficient of the treatment/control indicator in the above mixed model; Cohen's D = .064, 95% CI 2-sided [-.294 to .421], Standard Error of Mean .181 — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Consequences of Cannabis Use as Measured by the Marijuana Adolescent Consequences Questionnaire Using Dichotomous Response Scale as Previously Described Throughout This Trial Registration.
Description: Marijuana Adolescent Consequences Questionnaire will be used to assess past 3 month consequences of cannabis use. Consequences are measured by report of number of times incidents from the list of 26 items (e.g., quality of work suffered, had less energy, etc.) resulted from cannabis use. Responses will be dichotomized (0 = never, 1= greater than never) and summed for a total score reflecting total number of consequences.
  Response scale:
  Never 1-2 times 3-5 times 6-10 times More than 10 times
  Minimum score =0, maximum = 26. Higher score = more consequences.
Time Frame: 3-months post-baseline
Measure: Mean (Standard Deviation); unit: total number of consequences (count)
Arm/Group | Social Media Intervention | Control
Number analyzed (Participants) | 70 | 65
total number of consequences (count) | 10.1 (5.7) | 10.2 (5.7)
Statistical Analysis 1: Comparison: Social Media Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Other — Two-sided test of the null hypothesis of no difference between groups; p = .656, t-test, 2 sided; The p-value is for the coefficient of the treatment/control indicator in the above mixed model; Cohen's D = -.078, 95% CI 2-sided [-.425 to .269], Standard Error of Mean .175 — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: Consequences of Cannabis Use as Measured by the Marijuana Adolescent Consequences Questionnaire
Description: as for outcome 5
Time Frame: 6-months post-baseline
Measure: Mean (Standard Deviation); unit: total consequences (count)
Arm/Group | Social Media Intervention | Control
Number analyzed (Participants) | 68 | 65
total consequences (count) | 9.9 (6.5) | 8.8 (5.6)
Statistical Analysis 1: Comparison: Social Media Intervention vs Control; Test type: Other — Two-sided test of the null hypothesis of no difference between groups; p = .158, t-test, 2 sided — The p-value is for the coefficient of the treatment/control indicator in the above mixed model; Cohen's D = -.339, 95% CI 2-sided [-.746 to 0.067], Standard Error of Mean .205 — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Perceived Risk of Cannabis Use as Measured by 2 Modified Items From the Monitoring the Future Survey
Description: Two items rating current opinion on a scale from "no risk" to "great risk" of their perceived risk harm from occasional cannabis use and regular use.
  Items are--
  How much do you think people risk harming themselves (physically or in other ways), if they:
  1. Use marijuana or marijuana products occasionally
  2. Use marijuana or marijuana products regularly
  Response options are:
  1. No risk
  2. Slight risk
  3. Moderate risk
  4. Great risk
  Answers from both items are added together. The total range of two items summed can be 2-8. Higher totals indicate higher perceived risk.
Time Frame: 3-months post-baseline
Measure: Mean (Standard Deviation); unit: total of two items
Arm/Group | Social Media Intervention | Control
Number analyzed (Participants) | 70 | 65
total of two items | 3.1 (1.1) | 3.5 (1.1)
Statistical Analysis 1: Comparison: Social Media Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Other — Two-sided test of the null hypothesis of no difference between groups; p = .422, t-test, 2 sided; The p-value is for the coefficient of the treatment/control indicator in the above mixed model; Cohen's D = .143, 95% CI 2-sided [-.210 to .495], Standard Error of Mean .178 — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Perceived Risk of Cannabis Use as Measured by Modified Items From the Monitoring the Future Survey
Description: as for outcome 7
Time Frame: 6-months post-baseline
Measure: Mean (Standard Deviation); unit: total of two items
Arm/Group | Social Media Intervention | Control
Number analyzed (Participants) | 68 | 65
total of two items | 3.3 (1.2) | 3.5 (1.3)
Statistical Analysis 1: Comparison: Social Media Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Other — Two-sided test of the null hypothesis of no difference between groups; p = .882, t-test, 2 sided; Cohen's D = .027, 95% CI 2-sided [-.328 to .381], Standard Error of Mean .179 — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Peer Approval/Disapproval of Cannabis Use as Measured by Item Modified From Monitoring the Future Survey
Description: One item rating of current perception of whether their close friends would disapprove of their cannabis use (regardless of how much they use), rated as:
  1. Not disapprove
  2. Disapprove
  3. Strongly disapprove
Time Frame: 3 months post-baseline
Population: Number of participants analyzed is due to missing data
Measure: Mean (Standard Deviation); unit: score on the single item
Arm/Group | Social Media Intervention | Control
Number analyzed (Participants) | 70 | 64
score on the single item | 1.0 (0.2) | 1.0 (0.1)
Statistical Analysis 1: Comparison: Social Media Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Other — Two-sided test of the null hypothesis of no difference between groups; p = .497, t-test, 2 sided — The p-value is for the coefficient of the treatment/control indicator in the above mixed model; Cohen's D = -.197, 95% CI 2-sided [-.728 to .334], Standard Error of Mean .268 — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Peer Approval/Disapproval of Cannabis Use as Measured by Item Modified From Monitoring the Future Survey
Description: One item rating of current perception of whether their close friends would disapprove of their cannabis use (regardless of how much they use), rated as: 1 Not disapprove 2 Disapprove 3 Strongly disapprove
Time Frame: 6 months post-baseline
Population: Number of participants analyzed is due to missing data
Measure: Mean (Standard Deviation); unit: score on the single item
Arm/Group | Social Media Intervention | Control
Number analyzed (Participants) | 68 | 64
score on the single item | 1.1 (0.4) | 1.1 (0.3)
Statistical Analysis 1: Comparison: Social Media Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Other — Two-sided test of the null hypothesis of no difference between groups; p = .813, t-test, 2 sided — The p-value is for the coefficient of the treatment/control indicator in the above mixed model; Cohen's D = -.042, 95% CI 2-sided [-.398 to .313], Standard Error of Mean .180 — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Cannabis Impaired Driving as Measured by 5 Items From the Modified Young Adult Driving Questionnaire
Description: Five items from the modified Young Adult Driving Questionnaire will be used to assess past 3 month driving under the influence of cannabis. Response values will be summed for a total score.
  In the PAST 3 MONTHS...how many times did you drive within one hour after using marijuana or marijuana products containing THC?
  * how many times did you drive while a little high on marijuana or marijuana products containing THC?
  * how many times did you drive while very high on marijuana or marijuana products containing THC?
  * how many times did you drive when you knew your use of marijuana/marijuana products containing THC may already have affected your coordination?
  * how many times did you ride in a car or other vehicle driven by someone who had been using marijuana or marijuana products containing THC?
  Response options:
  0= Never
  1. Once
  2. Twice
  3. 3 times
  4. 4 times
  5. 5 times
  6. 6-9 times
  7. 10 or more times
Time Frame: 3 months post-baseline
Measure: Mean (Standard Deviation); unit: total of 5 items (range = 0 to 35)
Arm/Group | Social Media Intervention | Control
Number analyzed (Participants) | 70 | 65
total of 5 items (range = 0 to 35) | 10.2 (11.4) | 8.8 (10.4)
Statistical Analysis 1: Comparison: Social Media Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Other — Two-sided test of the null hypothesis of no difference between groups; p = .849, t-test, 2 sided — The p-value is for the coefficient of the treatment/control indicator in the above mixed model; Cohen's D = -.034, 95% CI 2-sided [-.381 to .314], Standard Error of Mean .176 — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Cannabis Impaired Driving as Measured by 5 Items From the Modified Young Adult Driving Questionnaire
Description: as for outcome 11
Time Frame: 6 months post-baseline
Measure: Mean (Standard Deviation); unit: total of 5 items (range 0 to 35)
Arm/Group | Social Media Intervention | Control
Number analyzed (Participants) | 68 | 65
total of 5 items (range 0 to 35) | 9.6 (11.1) | 7.2 (10.1)
Statistical Analysis 1: Comparison: Social Media Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Other — Two-sided test of the null hypothesis of no difference between groups; p = .667, t-test, 2 sided — The p-value is for the coefficient of the treatment/control indicator in the above mixed model; Cohen's D = -.118, 95% CI 2-sided [-.607 to .371], Standard Error of Mean .247 — The effect size used is the adjusted Cohen's D, calculated from the coefficient for treatment group in the mixed model, divided by total pooled SD (the square root of the sum of the residual variance+the variance of the group-level random effects

13. Secondary Outcome: Other Drug Use as Measured by Items Modified From Monitoring the Future Survey
Description: Items from the Monitoring the Future Survey will be used to assess past 30 day use of 6 other substances - substances used and number of times of use. Response values will be summed for a total score using mid-point of the range scoring.
  Substances assessed include: hallucinogens, opioids, stimulants, sedatives, lsd, ecstasy
  Response scale:
  0 0 Occasions
  1. 1-2 Occasions
  2. 3-5 Occasions
  3. 6-9 Occasions
  4. 10-19 Occasions
  5. 20-39 Occasions
  6. 40 or More Occasions
Time Frame: 3 months post-baseline
Measure: Mean (Standard Deviation); unit: total of 6 items using mid-point scoring
Arm/Group | Social Media Intervention | Control
Number analyzed (Participants) | 70 | 65
total of 6 items using mid-point scoring | 3.4 (7.9) | 1.0 (4.3)
Statistical Analysis 1: Comparison: Social Media Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Other — Two-sided test of the null hypothesis of no difference between groups; p = .051, t-test, 2 sided; The p-value is for the coefficient of the treatment/control indicator in the above mixed model; Cohen's D = -.342, 95% CI 2-sided [-.689 to .005], Standard Error of Mean .175 — [estimate comment as in outcome 12, analysis 1]

14. Secondary Outcome: Other Drug Use as Measured by Items Modified From Monitoring the Future Survey
Description: as for outcome 13
Time Frame: 6 months post-baseline
Measure: Mean (Standard Deviation); unit: total of 6 items using midpoint of range
Arm/Group | Social Media Intervention | Control
Number analyzed (Participants) | 68 | 65
total of 6 items using midpoint of range | 2.5 (7.2) | 1.9 (10.1)
Statistical Analysis 1: Comparison: Social Media Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Other — Two-sided test of the null hypothesis of no difference between groups; p = .714, t-test, 2 sided; The p-value is for the coefficient of the treatment/control indicator in the above mixed model; Cohen's D = -.064, 95% CI 2-sided [-.412 to .284], Standard Error of Mean .176; The effect size used is the adjusted Cohen's D, calculated from the coefficient for treatment group in the mixed model, divided by total pooled SD (the square root of the sum of the residual variance+the variance of the group-level random effects)

15. Secondary Outcome: Frequency of Alcohol Consumption as Reported on the Timeline Follow-Back (TLFB)
Description: 30-day TLFB self-report will be used to assess total number of days of alcohol consumption.
Time Frame: 3 months post-baseline
Population: Number of participants analyzed is due to focus on alcohol drinkers only
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Social Media Intervention | Control
Number analyzed (Participants) | 56 | 40
days | 6.0 (8.0) | 6.1 (8.1)
Statistical Analysis 1: Comparison: Social Media Intervention vs Control; : We fixed linear mixed effects models adjusted for baseline values, balancing factors (age, sex, recreational cannabis), and included a random intercept for group because this is an individually randomized group treatment trial. We tested for treatment effects with a two-sided test of the coefficient for the treatment/control indicator, and estimated Cohen's D (mean difference between the 2 groups at follow-up divided by the total variation not captured by the fixed effects) along with 95% CIs; Test type: Other — Two-sided test of the null hypothesis of no difference between groups; p = .603, t-test, 2 sided; The p-value is for the coefficient of the treatment/control indicator in the above mixed model; Cohen's D = -.110, 95% CI 2-sided [-.531 to .311], Standard Error of Mean .212 — [estimate comment as in outcome 1, analysis 1]

16. Secondary Outcome: Frequency of Alcohol Consumption as Reported on the Timeline Follow-Back (TLFB)
Description: 30-day TLFB self-report will be used to assess total number of days of alcohol consumption.
Time Frame: 6 months post-baseline
Population: Number of participants analyzed is due to focus on alcohol drinkers only
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Social Media Intervention | Control
Number analyzed (Participants) | 53 | 38
days | 4.9 (7.6) | 6.5 (7.8)
Statistical Analysis 1: Comparison: Social Media Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Other — Two-sided test of the null hypothesis of no difference between groups; p = .457, Cohen's D; The p-value is for the coefficient of the treatment/control indicator in the above mixed model; Cohen's D = .162, 95% CI 2-sided [-.273 to .597], Standard Error of Mean .219 — [estimate comment as in outcome 1, analysis 1]

17. Secondary Outcome: Quantity of Alcohol Consumption as Reported on the Timeline Follow-Back (TLFB)
Description: 30-day TLFB self-report will be used to assess the quantity of alcohol consumed.
Time Frame: 3 months post-baseline
Population: Number of participants analyzed is due to focus on alcohol drinkers only
Measure: Mean (Standard Deviation); unit: estimated standard drinks
Arm/Group | Social Media Intervention | Control
Number analyzed (Participants) | 56 | 40
estimated standard drinks | 17.1 (28.1) | 12.4 (15.4)
Statistical Analysis 1: Comparison: Social Media Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Other — Two-sided test of the null hypothesis of no difference between groups; p = .209, t-test, 2 sided; The p-value is for the coefficient of the treatment/control indicator in the above mixed model; Cohen's D = -.265, 95% CI 2-sided [-.686 to .156], Standard Error of Mean .212 — [estimate comment as in outcome 1, analysis 1]

18. Secondary Outcome: Quantity of Alcohol Consumption as Reported on the Timeline Follow-Back (TLFB)
Description: 30-day TLFB self-report will be used to assess the quantity of alcohol consumed.
Time Frame: 6 months post-baseline
Population: Number of participants analyzed is due to focus on alcohol drinkers only
Measure: Mean (Standard Deviation); unit: estimated standard drinks
Arm/Group | Social Media Intervention | Control
Number analyzed (Participants) | 38 | 53
estimated standard drinks | 14.3 (27.5) | 13.5 (15.8)
Statistical Analysis 1: Comparison: Social Media Intervention vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Other — Two-sided test of the null hypothesis of no difference between groups; p = .623, t-test, 2 sided; The p-value is for the coefficient of the treatment/control indicator in the above mixed model; Cohen's D = -.107, 95% CI 2-sided [-.541 to .328], Standard Error of Mean .219 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From baseline to 6-month follow-up. Note that adverse events were monitored but none occurred; this is a no more than minimal risk study.
Arm/Group | Social Media Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/73
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/73
Other Adverse Events (participants affected / at risk) | 0/76 | 0/73

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/89/NCT04187989/Prot_SAP_001.pdf
  • Informed Consent Form (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT04187989/ICF_000.pdf